CLINICAL TRIAL: NCT00490568
Title: An Open-label Extension to Study AVA102670 and AVA102672, to Assess the Long-term Safety and Efficacy of Rosiglitazone (Extended Release Tablets) as Adjunctive Therapy on Cognition in Subjects With Mild to Moderate Alzheimer's Disease.
Brief Title: Open-Label Extension Study Of Rosiglitazone XR As Adjunctive Therapy In Subjects With Mild-to-Moderate Alzheimers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on preliminary parent study results
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA102675
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-09

CONDITIONS: Alzheimer's Disease
Keywords: cognition; Alzheimer's disease; Rosiglitazone extended-release (XR); safety; adjunctive therapy; BRL-049653; tolerability; open-label extension
MeSH Terms: conditions — Alzheimer Disease

ARMS (1):
- Rosiglitazone XR (Experimental): Investigational drug
  Interventions: Drug: Rosiglitazone XR

INTERVENTIONS:
Drug: Rosiglitazone XR — Experimental drug

SUMMARY:
This is a Phase III, multicenter, open-label extension, single-group study in male and female outpatients with mild-to-moderate Alzheimer's disease (AD) who have completed either AVA102670 or AVA102672. All subjects will receive rosiglitazone extended-release (RSG XR) 4mg once daily for the first 4 weeks of the study followed by 8mg RSG XR as adjunctive therapy to their existing dose of acetylcholinesterase inhibitor. Subject participation will last until one of 5 conditions applies. After a 52-week open-label treatment phase, subjects will attend a final Follow-Up Visit 6 weeks after the end of treatment. The primary objective of this study is to evaluate the long-term safety and tolerability of RSG XR in subjects with mild-to-moderate AD who have completed either AVA102670 or AVA102672. The secondary objective of this study is to explore further the long-term efficacy of RSG XR in terms of cognitive function and overall clinical response as a function of apolipoprotein E (APOE) e4 allele status.

ELIGIBILITY:
Inclusion criteria:

* Successful completion of AVA102670 or AVA102672 without safety or tolerability issues. Regular caregiver.

Exclusion criteria:

* Congestive Heart Failure (NYHA 1-4), clinically significant peripheral edema, other neurological conditions that might disqualify participation. SAE, clinically significant laboratory abnormality or significant cardiovascular event during prior study.

Ages: 51 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1461 (Actual)
Dates: Start 2007-08-08 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (225):
- United States (41):
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Sherman Oaks, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, West Yarmouth, Massachusetts
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Stratford, New Jersey
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, South Ogden, Utah
  - GSK Investigational Site, Bennington, Vermont
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (6):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Godoy Cruz, Mendoza Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (10):
  - GSK Investigational Site, Hornsby, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Chermside, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Cheltenham, Victoria
  - GSK Investigational Site, Heidelberg Heights, Victoria
  - GSK Investigational Site, Kew, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Austria (2):
  - GSK Investigational Site, Hall in Tirol
  - GSK Investigational Site, Vienna
- Belgium (3):
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Woluwe-Saint-Lambert
- Bulgaria (2):
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (13):
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Kentville, Nova Scotia
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Whitby, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
  - GSK Investigational Site, Québec
- Chile (3):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Providencia / Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Czechia (4):
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Trutnov
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kuopio
- France (24):
  - GSK Investigational Site, Bourg-en-Bresse
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Ivry
  - GSK Investigational Site, La Seyne-sur-Mer
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Luynes
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Metz
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Rodez
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Saint-Ouen-la-Rouërie
  - GSK Investigational Site, Sautron
  - GSK Investigational Site, Tinténiac
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Vichy
- Germany (42):
  - GSK Investigational Site, Aalen, Baden-Wurttemberg
  - GSK Investigational Site, Ellwangen, Baden-Wurttemberg
  - GSK Investigational Site, Ludwigsburg, Baden-Wurttemberg
  - GSK Investigational Site, Ostfildern, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Alzenau in Unterfranken, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Bad Saarow, Brandenburg
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Erbach im Odenwald, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Bockhorn, Lower Saxony
  - GSK Investigational Site, Ganderkesee, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Lüneburg, Lower Saxony
  - GSK Investigational Site, Westerstede, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bad Honnef, North Rhine-Westphalia
  - GSK Investigational Site, Baesweiler, North Rhine-Westphalia
  - GSK Investigational Site, Bergisch Gladbach, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
  - GSK Investigational Site, Jülich, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Siegen, North Rhine-Westphalia
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Gera, Thuringia
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Melíssia
  - GSK Investigational Site, Thessaloniki
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin
- Hungary (2):
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Szeged
- India (5):
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Varanasi
- Italy (12):
  - GSK Investigational Site, Chieti Scalo, Abruzzo
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, San Felice A Cancello Caserta, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Rho, Lombardy
  - GSK Investigational Site, Torrette (AN), The Marches
  - GSK Investigational Site, Arezzo, Tuscany
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Pisa, Tuscany
- Mexico (2):
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México
- Netherlands (6):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Blaricum
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hilversum
  - GSK Investigational Site, The Hague
- GSK Investigational Site, Pasig, Philippines
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Mosina
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Warsaw
- Portugal (2):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
- Slovenia (2):
  - GSK Investigational Site, Ljubljana
  - GSK Investigational Site, Šempeter v Savinj. Dolini
- South Africa (7):
  - GSK Investigational Site, Loeventstein
  - GSK Investigational Site, Oakdale
  - GSK Investigational Site, Richards Bay
  - GSK Investigational Site, Rosebank
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Waverley, Bloemfontein
  - GSK Investigational Site, Willows, X14, Pretoria
- South Korea (2):
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
- Spain (10):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Tarrasa, Barcelona
  - GSK Investigational Site, Valencia
- Sweden (5):
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Kalix
  - GSK Investigational Site, Mölndal
  - GSK Investigational Site, Sundsvall
  - GSK Investigational Site, Umeå
- United Kingdom (4):
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, West of Scotland Science Park, Glasgow

REFERENCES:
- [Background] Harrington C, Sawchak S, Chiang C, Davies J, Donovan C, Saunders AM, Irizarry M, Jeter B, Zvartau-Hind M, van Dyck CH, Gold M. Rosiglitazone does not improve cognition or global function when used as adjunctive therapy to AChE inhibitors in mild-to-moderate Alzheimer's disease: two phase 3 studies. Curr Alzheimer Res. 2011 Aug;8(5):592-606. doi: 10.2174/156720511796391935. PMID 21592048
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: AVA102675 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVA102675 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVA102675 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVA102675 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVA102675 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVA102675 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVA102675 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A open-label extension study to evaluate the long-term safety and tolerability of rosiglitazone extended-release (RSG XR) tablets in participants with mild-to moderate Alzheimer's Disease conducted in a total of 29 countries across 267 centers from 08 August 2007 to 30 May 2009.
Pre-assignment Details: Approximately 1800 participants were planned to be enrolled however a total of 1461 participants (after completing parent studies AVA102670/AVA102672) were enrolled and received open-label RSG-XR tablets.
Groups:
- RSG XR: Eligible participants who completed studies AVA102670 or AVA102672 entered in this open-label extension study. Participants received open-label RSG XR throughout the treatment period as adjunctive therapy to their existing dose of Acetylcholinesterase Inhibitor (AChEI) for Alzheimer's disease treatment. Participants took one tablet of study medication daily in the morning with or without food. All participants received oral 4 milligram (mg) once daily RSG XR for the first 4 weeks of the study (only for the first 4 weeks of the study). The RSG XR dose was then increased to 8 mg once daily from Week 4 through Week 52. The dose of RSG XR was reduced to 2mg once daily if the 8 mg dose was not well tolerated. Participants were not permitted to titrate back to 8 mg RSG XR.
Period: Overall Study
Arm/Group | RSG XR
Started | 1461
Completed | 97
Not Completed | 1364
Not completed — Adverse Event | 116
Not completed — Lost to Follow-up | 13
Not completed — Protocol Violation | 45
Not completed — Withdrawal by Subject | 135
Not completed — Still in the study at termination | 974
Not completed — Other | 1
Not completed — Exclusion criteria met | 1
Not completed — Caregiver related | 20
Not completed — Abnormal ECG | 25
Not completed — Participant refused follow-up | 9
Not completed — Legal representative withdrew consent | 1
Not completed — Disease progression | 4
Not completed — Unmet inclusion-exclusion criteria | 5
Not completed — Investigator decision | 3
Not completed — Non-Compliance | 7
Not completed — Efficacy related | 3
Not completed — Participant died | 1
Not completed — Participant withdrawal due to surgery | 1

BASELINE CHARACTERISTICS:
Groups:
- RSG XR (AVA102675): Eligible participants who completed studies AVA102670 or AVA102672 entered in this open-label extension study. Participants received open-label RSG XR throughout the treatment period as adjunctive therapy to their existing dose of AChEI for Alzheimer's disease treatment. Participants took one tablet of study medication daily in the morning with or without food. All participants received 4 mg once daily RSG XR for the first 4 weeks of the study (only for the first 4 weeks of the study). The RSG XR dose was then increased to 8 mg once daily from Week 4 through Week 52. The dose of RSG XR was reduced to 2mg once daily if the 8 mg dose was not well tolerated. Participants were not permitted to titrate back to 8 mg RSG XR.
Arm/Group | RSG XR (AVA102675)
Number analyzed (Participants) | 1461
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.9 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 843
  Male | 618
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 52
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 1396
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Severity of AEs
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The severity of the AE'S was categorized as mild, moderate and severe. Number of participants reporting AEs during the on treatment phase of the study.
Time Frame: Up to 76 Weeks
Population: All Subjects (Full population), comprised of all participants who took at least one dose of open-label study medication.
Measure: Count of Participants; unit: Participants
Groups:
- RSG XR: Eligible participants who completed studies AVA102670 or AVA102672 entered in this open-label extension study. Participants received open-label RSG XR throughout the treatment period as adjunctive therapy to their existing dose of AChEI for Alzheimer's disease treatment. Participants took one tablet of study medication daily in the morning with or without food. All participants received 4 mg once daily RSG XR for the first 4 weeks of the study (only for the first 4 weeks of the study). The RSG XR dose was then increased to 8 mg once daily from Week 4 through Week 52. The dose of RSG XR was reduced to 2mg once daily if the 8 mg dose was not well tolerated. Participants were not permitted to titrate back to 8 mg RSG XR..
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Participants
  Any AE | 724
  Mild AE | 345
  Moderate AE | 289
  Severe AE | 88

2. Secondary Outcome: Number Participants With Serious Adverse Events (SAEs) and Deaths
Description: A SAE is defined as any untoward medical occurrence that, at any dose results in death, is a life-threatening condition, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, or a congenital anomaly or birth defect. Number of participants with SAEs and deaths were reported for treatment duration of the study.
Time Frame: Up to 76 Weeks
Population: All subject (Full population)
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Participants
  Any SAE | 126
  Deaths | 20

3. Secondary Outcome: Number of Participants With Adverse Event of Oedema
Description: Oedema was considered as adverse event of special interest (AESI). The process for AESI selection was based on RSG's pharmacologic class and relevant AEs potentially associated with RSG. The number of participants and their percentage for the adverse event of the various types of oedema were reported.
Time Frame: Up to 76 Weeks
Population: All subject (Full population)
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Participants
  Oedema peripheral | 130
  Face oedema | 8
  Pitting oedema | 5
  Oedema | 3
  Pulmonary oedema | 1
  Eyelid oedema | 1

4. Secondary Outcome: Change From Baseline in Vital Sign Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs SBP and DBP were measured at each visit. All measurements were made on the participant non-dominant arm supported at heart level, using the same cuff size and same equipment. Blood pressure was measured once, after the participant sat quietly for at least 5 minutes. DBP was measured at the disappearance of Korotkoff sounds (Phase V). If the participant was a smoker or used tobacco products, a period of 30 minutes without tobacco was allowed before taking these measurements. Baseline for the open-label study was the latest assessment from Week 48 of parent studies to the first dose of open-label medication. Change from Baseline was measured as the blood pressure value recorded at specified visit minus the Baseline value.
Time Frame: Up to 70 Weeks (including follow up)
Population: All subject (Full population). Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
millimeters of mercury (mmHg)
  SBP at Week 4: number analyzed (Participants) | 1395
  SBP at Week 4 | -1.4 (14.10)
  SBP at Week 8: number analyzed (Participants) | 1274
  SBP at Week 8 | -2.4 (14.73)
  SBP at Week 12: number analyzed (Participants) | 1146
  SBP at Week 12 | -2.7 (14.73)
  SBP at Week 16: number analyzed (Participants) | 1061
  SBP at Week 16 | -3.7 (15.02)
  SBP at Week 24: number analyzed (Participants) | 892
  SBP at Week 24 | -2.1 (15.51)
  SBP at Week 36: number analyzed (Participants) | 666
  SBP at Week 36 | -1.4 (15.14)
  SBP at Week 52: number analyzed (Participants) | 251
  SBP at Week 52 | -1.7 (16.18)
  SBP at Week 64: number analyzed (Participants) | 15
  SBP at Week 64 | -2.2 (13.78)
  SBP at Follow-up: number analyzed (Participants) | 1280
  SBP at Follow-up | -1.8 (15.60)
  DBP at Week 4: number analyzed (Participants) | 1395
  DBP at Week 4 | -1.4 (9.41)
  DBP at Week 8: number analyzed (Participants) | 1274
  DBP at Week 8 | -2.0 (9.53)
  DBP at Week 12: number analyzed (Participants) | 1146
  DBP at Week 12 | -2.1 (9.74)
  DBP at Week 16: number analyzed (Participants) | 1061
  DBP at Week 16 | -2.4 (9.62)
  DBP at Week 24: number analyzed (Participants) | 892
  DBP at Week 24 | -2.4 (9.48)
  DBP at Week 36: number analyzed (Participants) | 666
  DBP at Week 36 | -2.0 (9.85)
  DBP at Week 52: number analyzed (Participants) | 251
  DBP at Week 52 | -3.6 (9.94)
  DBP at Week 64: number analyzed (Participants) | 15
  DBP at Week 64 | -6.3 (6.72)
  DBP at Follow-up: number analyzed (Participants) | 1280
  DBP at Follow-up | -0.9 (10.23)

5. Secondary Outcome: Change From Baseline in Vital Sign Heart Rate (HR)
Description: Vital sign HR was measured at each visit. HR was measured once, after the participant sat quietly for at least 5 minutes. Baseline for the open-label study was the latest assessment from Week 48 of parent studies to the first dose of open-label medication. Change from Baseline was measured as the HR at specified visit minus the Baseline value.
Time Frame: Up to 70 Weeks (including follow up)
Population: All subject (Full population). Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
beats per minute (bpm)
  HR at Week 4: number analyzed (Participants) | 1391
  HR at Week 4 | 1.0 (8.95)
  HR at Week 8: number analyzed (Participants) | 1271
  HR at Week 8 | 1.8 (9.60)
  HR at Week 12: number analyzed (Participants) | 1142
  HR at Week 12 | 1.6 (9.77)
  HR at Week 16: number analyzed (Participants) | 1061
  HR at Week 16 | 1.6 (9.66)
  HR at Week 24: number analyzed (Participants) | 888
  HR at Week 24 | 0.9 (9.99)
  HR at Week 36: number analyzed (Participants) | 665
  HR at Week 36 | 1.3 (9.86)
  HR at Week 52: number analyzed (Participants) | 251
  HR at Week 52 | 0.7 (8.54)
  HR at Week 64: number analyzed (Participants) | 15
  HR at Week 64 | 1.0 (8.02)
  HR at Follow-up: number analyzed (Participants) | 1276
  HR at Follow-up | 0.9 (10.03)

6. Secondary Outcome: Change From Baseline in Vital Sign Body Weight (BW)
Description: BW was measured at all visits, without shoes and wearing light clothing. Baseline for the open-label study was the latest assessment from Week 48 of parent studies to the first dose of open-label medication. Change from Baseline was measured as the body weight at specified visit minus the Baseline value.
Time Frame: Up to 70 Weeks (including follow up)
Population: All subject (Full population). Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
kg
  BW at Week 4: number analyzed (Participants) | 1391
  BW at Week 4 | 0.3 (2.04)
  BW at Week 8: number analyzed (Participants) | 1263
  BW at Week 8 | 0.6 (2.45)
  BW at Week 12: number analyzed (Participants) | 1139
  BW at Week 12 | 0.6 (2.43)
  BW at Week 16: number analyzed (Participants) | 1057
  BW at Week 16 | 0.7 (3.53)
  BW at Week 24: number analyzed (Participants) | 889
  BW at Week 24 | 0.6 (2.95)
  BW at Week 36: number analyzed (Participants) | 666
  BW at Week 36 | 1.0 (4.08)
  BW at Week 52: number analyzed (Participants) | 251
  BW at Week 52 | 1.2 (3.82)
  BW at Week 64: number analyzed (Participants) | 15
  BW at Week 64 | 1.4 (2.52)
  BW at Follow-up: number analyzed (Participants) | 1268
  BW at Follow-up | 0.5 (3.15)

7. Secondary Outcome: Change From Baseline in Non-fasting Measures of Lipid Metabolism Namely Total Cholesterol (TC), High Density Lipoprotein (HDL), Low Density Lipoprotein (LDL), Triglycerides
Description: The clinical chemistry data included non-fasting measures of lipid metabolism (TC,HDL,LDL,triglycerides). Baseline for the open-label study was the latest assessment from Week 48 of parent studies to the first dose of open-label medication. Change from Baseline was measured as the lipids (TC,HDL,LDL,triglycerides) value recorded at specified visit minus the Baseline value.
Time Frame: Up to 82 Weeks (including follow up)
Population: All subject (Full population). Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimole per litre (mmol/l)
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
millimole per litre (mmol/l)
  TC at Week 4: number analyzed (Participants) | 1313
  TC at Week 4 | 0.076 (0.6828)
  TC at Week 16: number analyzed (Participants) | 1038
  TC at Week 16 | 0.201 (0.8666)
  TC at Week 36: number analyzed (Participants) | 639
  TC at Week 36 | 0.246 (0.9649)
  TC at Week 52: number analyzed (Participants) | 234
  TC at Week 52 | 0.174 (1.1437)
  TC at Week 76: number analyzed (Participants) | 2
  TC at Week 76 | -0.715 (0.3041)
  TC at follow up: number analyzed (Participants) | 888
  TC at follow up | 0.093 (0.9377)
  HDL at Week 4: number analyzed (Participants) | 1313
  HDL at Week 4 | 0.007 (0.2008)
  HDL at Week 16: number analyzed (Participants) | 1036
  HDL at Week 16 | -0.014 (0.2427)
  HDL at Week 36: number analyzed (Participants) | 639
  HDL at Week 36 | -0.026 (0.2487)
  HDL at Week 52: number analyzed (Participants) | 234
  HDL at Week 52 | -0.035 (0.2512)
  HDL at Week 76: number analyzed (Participants) | 1
  HDL at Week 76 | 0.050 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  HDL at follow up: number analyzed (Participants) | 887
  HDL at follow up | -0.058 (0.2605)
  LDL at Week 4: number analyzed (Participants) | 1263
  LDL at Week 4 | 0.062 (0.6207)
  LDL at Week 16: number analyzed (Participants) | 1008
  LDL at Week 16 | 0.210 (0.7782)
  LDL at Week 36: number analyzed (Participants) | 623
  LDL at Week 36 | 0.281 (0.8863)
  LDL at Week 52: number analyzed (Participants) | 226
  LDL at Week 52 | 0.228 (1.0563)
  LDL at Week 76: number analyzed (Participants) | 1
  LDL at Week 76 | -0.200 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  LDL at follow up: number analyzed (Participants) | 853
  LDL at follow up | 0.148 (0.8336)
  Triglycerides at Week 4: number analyzed (Participants) | 1313
  Triglycerides at Week 4 | 0.004 (0.7845)
  Triglycerides at Week 16: number analyzed (Participants) | 1038
  Triglycerides at Week 16 | -0.025 (0.8053)
  Triglycerides at Week 36: number analyzed (Participants) | 639
  Triglycerides at Week 36 | -0.062 (0.8053)
  Triglycerides at Week 52: number analyzed (Participants) | 234
  Triglycerides at Week 52 | -0.092 (0.8521)
  Triglycerides at Week 76: number analyzed (Participants) | 2
  Triglycerides at Week 76 | -0.150 (0.9758)
  Triglycerides at follow up: number analyzed (Participants) | 888
  Triglycerides at follow up | -0.035 (0.8295)

8. Secondary Outcome: Number of Participants With SBP and DBP Values of Potential Clinical Concern (PCC)
Description: The frequency of participant vital sign sitting blood pressure was obtained to check if the values lie outside of a pre-determined reference range (RR) for SBP 90-140 mmHg, DBP 50-90 mmHg or have a change from Baseline of PCC for SBP increase from Baseline (IFB) >=40, decrease from Baseline (DFB) >= 30 for and for DBP (IFB) >= 30 ,DFB >= 20. The number of participants with values of PCC at any time on treatment (ATOT) and follow up were reported.
Time Frame: Up to 70 Weeks (including follow up)
Population: All subject (Full population). Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Participants
  ATOT,SBP(RR)>140 or <90: number analyzed (Participants) | 1409
  ATOT,SBP(RR)>140 or <90 | 520
  ATOT,SBP(IFB)>=40: number analyzed (Participants) | 1409
  ATOT,SBP(IFB)>=40 | 33
  ATOT,SBP(DFB)>=30: number analyzed (Participants) | 1409
  ATOT,SBP(DFB)>=30 | 179
  Follow up,SBP(RR)>140 or <90: number analyzed (Participants) | 1280
  Follow up,SBP(RR)>140 or <90 | 240
  Follow up,SBP(IFB)>=40: number analyzed (Participants) | 1280
  Follow up,SBP(IFB)>=40 | 13
  Follow up,SBP(DFB)>=30: number analyzed (Participants) | 1280
  Follow up,SBP(DFB)>=30 | 63
  ATOT,DBP(RR)>90 or<50: number analyzed (Participants) | 1409
  ATOT,DBP(RR)>90 or<50 | 141
  ATOT,DBP(IFB)>=30: number analyzed (Participants) | 1409
  ATOT,DBP(IFB)>=30 | 20
  ATOT,DBP(DFB)>= 20: number analyzed (Participants) | 1409
  ATOT,DBP(DFB)>= 20 | 211
  Follow up,DBP(RR)>90 or<50: number analyzed (Participants) | 1280
  Follow up,DBP(RR)>90 or<50 | 54
  Follow up,DBP(IFB)>=30: number analyzed (Participants) | 1280
  Follow up,DBP(IFB)>=30 | 5
  Follow up, DBP(DFB)>= 20: number analyzed (Participants) | 1280
  Follow up, DBP(DFB)>= 20 | 67

9. Secondary Outcome: Number of Participants With HR Values of PCC ATOT
Description: HR was measured once, after the participant sat quietly for at least 5 minutes. The frequency of participant vital sign heart rate was obtained to check if the values lie outside of a pre-determined reference range (RR) 50-100 bpm or have a change from Baseline of PCC IFB >=30 and DFB >=30. The number of participants with values of PCC including follow up were reported.
Time Frame: Up to 70 Weeks (including follow up)
Population: All subject (Full population). Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Participants
  ATOT,HR (RR)>100 or <50: number analyzed (Participants) | 1409
  ATOT,HR (RR)>100 or <50 | 55
  ATOT,HR (IFB)>=30: number analyzed (Participants) | 1409
  ATOT,HR (IFB)>=30 | 25
  ATOT,HR (DFB)>=30: number analyzed (Participants) | 1409
  ATOT,HR (DFB)>=30 | 14
  Follow up,HR (RR)>100 or <50: number analyzed (Participants) | 1276
  Follow up,HR (RR)>100 or <50 | 18
  Follow up,HR (IFB)>=30: number analyzed (Participants) | 1276
  Follow up,HR (IFB)>=30 | 11
  Follow up,HR (DFB)>=30: number analyzed (Participants) | 1276
  Follow up,HR (DFB)>=30 | 6

10. Secondary Outcome: Number of Participants With BW Values of PCC ATOT
Description: The frequency of participant vital sign weight was obtained to check if the values have CFB of PCC IFB >=7 percent. With the exception of Week 4, when participants were first titrated to the 8mg RSG XR dose, at every time point in the study where weight was measured the percentage of participants experienced an increase in BW of PCC was approximately 2 times greater than the percentage of participants experiencing an decrease in BW of PCC DFB >=7 percent. The number of participants with values of PCC including follow up were reported.
Time Frame: Up to 70 Weeks (including follow up)
Population: All subject (Full population). Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Participants
  ATOT, BW(IFB)>=7 percent: number analyzed (Participants) | 1408
  ATOT, BW(IFB)>=7 percent | 188
  ATOT, BW(DFB)>= 7 percent: number analyzed (Participants) | 1408
  ATOT, BW(DFB)>= 7 percent | 83
  Follow up, BW(IFB)>=7 percent: number analyzed (Participants) | 1270
  Follow up, BW(IFB)>=7 percent | 90
  Follow up, BW(DFB)>= 7 percent: number analyzed (Participants) | 1270
  Follow up, BW(DFB)>= 7 percent | 51

11. Secondary Outcome: Number of Participants With Hematology Parameters of PCC ATOT
Description: The hematology data included eosinophils, haematocrit, haemoglobin, lymphocytes, mean corpuscular haemoglobin (MCH), mean corpuscular volume (MCV), monocytes, platelet count, red cell distribution width (RDW), red blood cell (RBC) count, segmented neutrophils (SN), total neutrophils (TN), white blood cell (WBC) count. The number of participants with values of PCC (defined as high and low) ATOT were reported.
Time Frame: Up to Week 82 (including follow up)
Population: All subject (Full population). Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Participants
  ATOT, Eosinophils (high): number analyzed (Participants) | 1384
  ATOT, Eosinophils (high) | 2
  ATOT, Haematocrit (low): number analyzed (Participants) | 1385
  ATOT, Haematocrit (low) | 8
  Follow up, Haematocrit (low): number analyzed (Participants) | 910
  Follow up, Haematocrit (low) | 6
  ATOT, Haemoglobin (high): number analyzed (Participants) | 1385
  ATOT, Haemoglobin (high) | 2
  ATOT, Haemoglobin (low): number analyzed (Participants) | 1385
  ATOT, Haemoglobin (low) | 74
  Follow up, Hemoglobin (high): number analyzed (Participants) | 910
  Follow up, Hemoglobin (high) | 2
  Follow up, Hemoglobin (low): number analyzed (Participants) | 910
  Follow up, Hemoglobin (low) | 25
  ATOT, Lymphocytes (high): number analyzed (Participants) | 1384
  ATOT, Lymphocytes (high) | 3
  ATOT, Lymphocytes (low): number analyzed (Participants) | 1384
  ATOT, Lymphocytes (low) | 21
  Follow up, Lymphocytes (high): number analyzed (Participants) | 909
  Follow up, Lymphocytes (high) | 3
  Follow up, Lymphocytes (low): number analyzed (Participants) | 909
  Follow up, Lymphocytes (low) | 9
  ATOT, MCH (low): number analyzed (Participants) | 1211
  ATOT, MCH (low) | 5
  Follow up, MCH (low): number analyzed (Participants) | 785
  Follow up, MCH (low) | 1
  ATOT, MCV (low): number analyzed (Participants) | 1385
  ATOT, MCV (low) | 1
  ATOT, monocytes (high): number analyzed (Participants) | 1384
  ATOT, monocytes (high) | 1
  ATOT, monocytes (low): number analyzed (Participants) | 1384
  ATOT, monocytes (low) | 61
  Follow up, monocytes (low): number analyzed (Participants) | 909
  Follow up, monocytes (low) | 23
  ATOT, platelet count (high): number analyzed (Participants) | 1381
  ATOT, platelet count (high) | 7
  ATOT, platelet count (low): number analyzed (Participants) | 1381
  ATOT, platelet count (low) | 5
  ATOT, RDW (high): number analyzed (Participants) | 1385
  ATOT, RDW (high) | 158
  Follow up, RDW (high): number analyzed (Participants) | 910
  Follow up, RDW (high) | 45
  ATOT, RBC (low): number analyzed (Participants) | 1385
  ATOT, RBC (low) | 12
  Follow up, RBC (low): number analyzed (Participants) | 910
  Follow up, RBC (low) | 4
  ATOT, SN (high): number analyzed (Participants) | 1384
  ATOT, SN (high) | 6
  ATOT, SN (low): number analyzed (Participants) | 1384
  ATOT, SN (low) | 15
  Follow up, SN (high): number analyzed (Participants) | 909
  Follow up, SN (high) | 3
  Follow up, SN (low): number analyzed (Participants) | 909
  Follow up, SN (low) | 3
  ATOT, TN (high): number analyzed (Participants) | 1384
  ATOT, TN (high) | 3
  ATOT, TN (low): number analyzed (Participants) | 1384
  ATOT, TN (low) | 15
  Follow up, TN (high): number analyzed (Participants) | 909
  Follow up, TN (high) | 2
  Follow up, TN (low): number analyzed (Participants) | 909
  Follow up, TN (low) | 3
  ATOT, WBC (high): number analyzed (Participants) | 1384
  ATOT, WBC (high) | 5
  ATOT, WBC (low): number analyzed (Participants) | 1384
  ATOT, WBC (low) | 22
  Follow up, WBC (high): number analyzed (Participants) | 909
  Follow up, WBC (high) | 3
  Follow up, WBC (low): number analyzed (Participants) | 909
  Follow up, WBC (low) | 11

12. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters (Including Lipids) of PCC ATOT
Description: The clinical chemistry data included alanine amino transferase (ALT), albumin, aldolase, asparatate amino transferase (AST), BUN/creatinine ratio, carbon dioxide(CO2) content, chloride, cholesterol, creatinine kinase (CK), creatinine, direct bilirubin (DB), gamma glutamyl transferase (GGT), glucose, glycosylated Hemoglobin (HbA1C), HDL, LDL, lactate dehydrogenase (LD), magnesium, potassium, sodium, total bilirubin (TB), triglycerides, troponin I, urea. The number of participants with values of PCC (defined as high and low) ATOT were reported.
Time Frame: Up to Week 82 (including follow up)
Population: All subject population (Full population). Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Participants
  Follow up, ALT (high): number analyzed (Participants) | 908
  Follow up, ALT (high) | 2
  Follow up, Albumin (low): number analyzed (Participants) | 909
  Follow up, Albumin (low) | 1
  ATOT, Aldolase (high): number analyzed (Participants) | 464
  ATOT, Aldolase (high) | 16
  ATOT, Aldolase (low): number analyzed (Participants) | 464
  ATOT, Aldolase (low) | 78
  Follow up, Aldolase (high): number analyzed (Participants) | 146
  Follow up, Aldolase (high) | 3
  Follow up, Aldolase (low): number analyzed (Participants) | 146
  Follow up, Aldolase (low) | 14
  ATOT, AST (high): number analyzed (Participants) | 1385
  ATOT, AST (high) | 2
  Follow up, AST (high): number analyzed (Participants) | 908
  Follow up, AST (high) | 3
  ATOT, BUN/creatinine ratio (high): number analyzed (Participants) | 1385
  ATOT, BUN/creatinine ratio (high) | 87
  Follow up, BUN/creatinine ratio (high): number analyzed (Participants) | 908
  Follow up, BUN/creatinine ratio (high) | 37
  ATOT, CO2 content (low): number analyzed (Participants) | 1384
  ATOT, CO2 content (low) | 2
  Follow up, CO2 content (low): number analyzed (Participants) | 908
  Follow up, CO2 content (low) | 3
  ATOT, chloride (high): number analyzed (Participants) | 1385
  ATOT, chloride (high) | 1
  ATOT, cholesterol (high): number analyzed (Participants) | 1383
  ATOT, cholesterol (high) | 175
  Follow up, cholesterol (high): number analyzed (Participants) | 907
  Follow up, cholesterol (high) | 50
  ATOT, CK (high): number analyzed (Participants) | 1385
  ATOT, CK (high) | 131
  Follow up, CK (high): number analyzed (Participants) | 908
  Follow up, CK (high) | 40
  ATOT, Creatinine (high): number analyzed (Participants) | 1385
  ATOT, Creatinine (high) | 27
  Follow up, creatinine (high): number analyzed (Participants) | 908
  Follow up, creatinine (high) | 10
  ATOT, DB (high): number analyzed (Participants) | 1385
  ATOT, DB (high) | 4
  ATOT, GGT (high): number analyzed (Participants) | 1385
  ATOT, GGT (high) | 7
  Follow up, GGT (high): number analyzed (Participants) | 908
  Follow up, GGT (high) | 2
  ATOT, Glucose (high): number analyzed (Participants) | 1385
  ATOT, Glucose (high) | 100
  ATOT, Glucose (low): number analyzed (Participants) | 1385
  ATOT, Glucose (low) | 40
  Follow up, glucose (high): number analyzed (Participants) | 908
  Follow up, glucose (high) | 31
  Follow up, glucose (low): number analyzed (Participants) | 908
  Follow up, glucose (low) | 13
  ATOT, HbA1c (high): number analyzed (Participants) | 742
  ATOT, HbA1c (high) | 2
  ATOT, HDL (low): number analyzed (Participants) | 1383
  ATOT, HDL (low) | 11
  Follow up, HDL (low): number analyzed (Participants) | 906
  Follow up, HDL (low) | 7
  ATOT, LDL (low): number analyzed (Participants) | 1368
  ATOT, LDL (low) | 469
  Follow up, LDL (low): number analyzed (Participants) | 888
  Follow up, LDL (low) | 211
  ATOT, LD (high): number analyzed (Participants) | 1384
  ATOT, LD (high) | 1
  Follow up, LD (high): number analyzed (Participants) | 909
  Follow up, LD (high) | 1
  ATOT, Magnesium (low): number analyzed (Participants) | 1385
  ATOT, Magnesium (low) | 1
  Follow up, Magnesium (low): number analyzed (Participants) | 909
  Follow up, Magnesium (low) | 1
  ATOT, Potassium (high): number analyzed (Participants) | 1384
  ATOT, Potassium (high) | 17
  ATOT, Potassium (low): number analyzed (Participants) | 1384
  ATOT, Potassium (low) | 1
  Follow up, Potassium (high): number analyzed (Participants) | 909
  Follow up, Potassium (high) | 2
  Follow up, Potassium (low): number analyzed (Participants) | 909
  Follow up, Potassium (low) | 1
  ATOT, Sodium (high): number analyzed (Participants) | 1385
  ATOT, Sodium (high) | 2
  ATOT, Sodium (low): number analyzed (Participants) | 1385
  ATOT, Sodium (low) | 4
  Follow up, Sodium (low): number analyzed (Participants) | 909
  Follow up, Sodium (low) | 1
  ATOT, TB (high): number analyzed (Participants) | 1386
  ATOT, TB (high) | 1
  Follow up, TB (high): number analyzed (Participants) | 908
  Follow up, TB (high) | 1
  ATOT, Triglycerides (high): number analyzed (Participants) | 1383
  ATOT, Triglycerides (high) | 1
  ATOT, Troponin I (high): number analyzed (Participants) | 426
  ATOT, Troponin I (high) | 13
  Follow up, Troponin I (high): number analyzed (Participants) | 142
  Follow up, Troponin I (high) | 2
  ATOT, Urea (high): number analyzed (Participants) | 1385
  ATOT, Urea (high) | 97
  Follow up, Urea (high): number analyzed (Participants) | 909
  Follow up, Urea (high) | 42

13. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive (ADAS-cog) Total Score as a Function of Apolipoprotein E (APOE) ε4 Status.
Description: The 11-item ADAS-Cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. Scores ranged from 0 to 70 with higher scores indicating greater dysfunction. Baseline for the open-label study was the latest assessment from Week 48 of parent studies to the first dose of open-label medication (Week 0). Change from Baseline was calculated as the Baseline value minus the value at the specified time point.
Time Frame: Baseline (Week 0) and Week 24, 52
Population: All subject (Full population). Only those participants available at the specified time points were analyzed. The analysis was done on the full population and was repeated for APOE subgroups (negative, positive, homozygotes, heterozygotes).
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Scores on scale
  Week 24 (Full population): number analyzed (Participants) | 973
  Week 24 (Full population) | 2.5 (5.51)
  Week 52 (Full population): number analyzed (Participants) | 308
  Week 52 (Full population) | 5.1 (6.82)
  Week 24 (APOE4 negatives): number analyzed (Participants) | 404
  Week 24 (APOE4 negatives) | 2.3 (5.28)
  Week 52 (APOE4 negatives): number analyzed (Participants) | 135
  Week 52 (APOE4 negatives) | 4.8 (6.44)
  Week 24 (APOE4 positives): number analyzed (Participants) | 569
  Week 24 (APOE4 positives) | 2.6 (5.66)
  Week 52(APOE4 positives): number analyzed (Participants) | 173
  Week 52(APOE4 positives) | 5.4 (7.11)
  Week 24 (APOE4 E4 homozygotes): number analyzed (Participants) | 126
  Week 24 (APOE4 E4 homozygotes) | 2.7 (5.77)
  Week 52 (APOE4 E4 homozygotes): number analyzed (Participants) | 39
  Week 52 (APOE4 E4 homozygotes) | 5.2 (7.49)
  Week 24 (APOE4 E4 heterozygotes): number analyzed (Participants) | 443
  Week 24 (APOE4 E4 heterozygotes) | 2.6 (5.63)
  Week 52 (APOE4 E4 heterozygotes): number analyzed (Participants) | 134
  Week 52 (APOE4 E4 heterozygotes) | 5.4 (7.02)

14. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) Score as a Function of APOE ε4 Status.
Description: The CDR-SB is a validated clinical assessment of global function in par. with Alzheimer's disease (AD). Impairment was scored in each of 6 cognitive categories on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2, and severe = 3. The 6 individual category ratings, or box scores, were added together to give the CDR-Sum of Boxes which ranged from 0 to 18 (severe impairment). Baseline for the open-label study was the latest assessment from Week 48 of parent studies to the first dose of open-label medication (Week 0). Change from Baseline was calculated as the Baseline value minus the value at the specified time point.
Time Frame: Baseline (Week 0) and Week 24, 52
Population: All subject population. Only those participants available at the specified time points were analyzed. The analysis was done on the full population and was repeated for APOE subgroups (negatives, positives, homozygotes, heterozygotes).
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Scores on scale
  Week 24 (Full population): number analyzed (Participants) | 988
  Week 24 (Full population) | 0.7 (1.84)
  Week 52 (Full population): number analyzed (Participants) | 313
  Week 52 (Full population) | 1.6 (2.26)
  Week 24 (APOE4 negatives): number analyzed (Participants) | 409
  Week 24 (APOE4 negatives) | 0.6 (1.76)
  Week 52 (APOE4 negatives): number analyzed (Participants) | 139
  Week 52 (APOE4 negatives) | 1.3 (2.19)
  Week 24 (APOE4 positives): number analyzed (Participants) | 579
  Week 24 (APOE4 positives) | 0.7 (1.89)
  Week 52 (APOE4 positives): number analyzed (Participants) | 174
  Week 52 (APOE4 positives) | 1.9 (2.30)
  Week 24 (APOE4 E4 homozygotes): number analyzed (Participants) | 127
  Week 24 (APOE4 E4 homozygotes) | 0.9 (1.90)
  Week 52 (APOE4 E4 homozygotes): number analyzed (Participants) | 39
  Week 52 (APOE4 E4 homozygotes) | 1.9 (2.32)
  Week 24 (APOE4 E4 heterozygotes): number analyzed (Participants) | 452
  Week 24 (APOE4 E4 heterozygotes) | 0.7 (1.89)
  Week 52 (APOE4 E4 heterozygotes): number analyzed (Participants) | 135
  Week 52 (APOE4 E4 heterozygotes) | 1.9 (2.30)

15. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score as a Function of APOE ε4 Status.
Description: The MMSE consisted of 11 tests of orientation, memory (recent and immediate), concentration, language and praxis. Scores ranged from 0 to 30, with lower scores indicating greater cognitive impairment. Baseline for the open-label study was the latest assessment from Week 48 of parent studies to the first dose of open-label medication (Week 0). Change from Baseline was calculated as the Baseline value minus the value at the specified time point.
Time Frame: Baseline (Week 0) and Week 24, 52
Population: All subject (Full population). Only those participants available at the specified time points were analyzed. The analysis was done on the full population and was repeated for APOE subgroups (negatives, positives, homozygotes, heterozygotes).
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Scores on scale
  Week 24 (Full population): number analyzed (Participants) | 833
  Week 24 (Full population) | -1.2 (2.84)
  Week 52 (Full population): number analyzed (Participants) | 184
  Week 52 (Full population) | -2.3 (3.39)
  Week 24 (APOE4 negatives): number analyzed (Participants) | 353
  Week 24 (APOE4 negatives) | -0.7 (2.74)
  Week 52 (APOE4 negatives): number analyzed (Participants) | 77
  Week 52 (APOE4 negatives) | -1.5 (3.56)
  Week 24 (APOE4 positives): number analyzed (Participants) | 480
  Week 24 (APOE4 positives) | -1.5 (2.87)
  Week 52 (APOE4 positives): number analyzed (Participants) | 107
  Week 52 (APOE4 positives) | -2.8 (3.17)
  Week 24 (APOE4 E4 homozygotes): number analyzed (Participants) | 104
  Week 24 (APOE4 E4 homozygotes) | -1.5 (3.07)
  Week 52 (APOE4 E4 homozygotes): number analyzed (Participants) | 23
  Week 52 (APOE4 E4 homozygotes) | -2.5 (3.16)
  Week 24 (APOE4 E4 heterozygotes): number analyzed (Participants) | 376
  Week 24 (APOE4 E4 heterozygotes) | -1.5 (2.82)
  Week 52 (APOE4 E4 heterozygotes): number analyzed (Participants) | 84
  Week 52 (APOE4 E4 heterozygotes) | -2.9 (3.18)

16. Secondary Outcome: Change From Baseline in Disability Assessment for Dementia Scale (DAD) Total Score as a Function of APOE ε4 Status.
Description: DAD, assessed the ability of a participant to execute basic and instrumental activities of daily living (ADL) and leisure activities. The scale consists of 40 questions assessing basic and instrumental ADLs. This scale assesses a participant's ability to initiate, plan, and perform activities related to hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. Each item was scored as yes: 1, no: 0 and N/A: not applicable. Higher scores indicate less disability with a score of 100 indicating no disability and 0 indicating no functional ability. The percentage score was calculated as (DAD total score/total number of applicable items) * 100. Baseline for the open-label study was the latest assessment from Week 48 of parent studies to the first dose of open-label medication (Week 0). Change from Baseline was calculated as the Baseline value minus the value at the specified time point.
Time Frame: Baseline (Week 0) and Week 24, 52
Population: All subject (Full population). Only those participants available at the specified time points were analyzed.The analysis was done on the full population and was repeated for APOE subgroups (negatives, positives, homozygotes, heterozygotes).
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Scores on scale
  Week 24 (Full population): number analyzed (Participants) | 837
  Week 24 (Full population) | -5.6 (12.36)
  Week 52 (Full population): number analyzed (Participants) | 183
  Week 52 (Full population) | -10.8 (15.07)
  Week 24 (APOE4 negatives): number analyzed (Participants) | 354
  Week 24 (APOE4 negatives) | -4.6 (11.57)
  Week 52 (APOE4 negatives): number analyzed (Participants) | 77
  Week 52 (APOE4 negatives) | -10.9 (14.90)
  Week 24 (APOE4 positives): number analyzed (Participants) | 483
  Week 24 (APOE4 positives) | -6.2 (12.88)
  Week 52 (APOE4 positives): number analyzed (Participants) | 106
  Week 52 (APOE4 positives) | -10.7 (15.26)
  Week 24 (APOE4 E4 homozygotes): number analyzed (Participants) | 106
  Week 24 (APOE4 E4 homozygotes) | -5.6 (12.16)
  Week 52 (APOE4 E4 homozygotes): number analyzed (Participants) | 24
  Week 52 (APOE4 E4 homozygotes) | -12.6 (11.84)
  Week 24 (APOE4 E4 heterozygotes): number analyzed (Participants) | 377
  Week 24 (APOE4 E4 heterozygotes) | -6.4 (13.08)
  Week 52 (APOE4 E4 heterozygotes): number analyzed (Participants) | 82
  Week 52 (APOE4 E4 heterozygotes) | -10.1 (16.14)

17. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score as a Function of APOE ε4 Status.
Description: 12-domain caregiver assessment of behavioral disturbances occurring in dementia: delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability, motor disturbance, appetite, nighttime behavior. A screening question is asked about each sub-domain. If the responses to these questions=participant has problems with a particular sub-domain of behavior, the caregiver asked all the questions about that domain, rating the frequency (1=occasionally to 4=very frequently) on a 4-point scale, their severity (1=Mild to 3=Severe) on a 3-point scale, and the distress on a 5-point scale. Total score=sum of each domain score(range 0-144);higher score=greater behavioral disturbances. Baseline for the open-label study was the latest assessment from Week 48 of parent studies to the first dose of open-label medication (Week 0). Change from Baseline was calculated as the Baseline value minus the value at the specified time point.
Time Frame: Baseline (Week 0) and Week 24, 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | RSG XR
Number analyzed (Participants) | 1461
Score on scale
  Week 24 (Full population): number analyzed (Participants) | 835
  Week 24 (Full population) | 1.4 (7.87)
  Week 52 (Full population): number analyzed (Participants) | 183
  Week 52 (Full population) | 3.2 (10.90)
  Week 24 (APOE4 negatives): number analyzed (Participants) | 353
  Week 24 (APOE4 negatives) | 1.0 (7.26)
  Week 52 (APOE4 negatives): number analyzed (Participants) | 77
  Week 52 (APOE4 negatives) | 2.4 (7.74)
  Week 24 (APOE4 positives): number analyzed (Participants) | 482
  Week 24 (APOE4 positives) | 1.7 (8.29)
  Week 52 (APOE4 positives): number analyzed (Participants) | 106
  Week 52 (APOE4 positives) | 3.8 (12.71)
  Week 24 (APOE4 E4 homozygotes): number analyzed (Participants) | 105
  Week 24 (APOE4 E4 homozygotes) | 1.8 (7.75)
  Week 52 (APOE4 E4 homozygotes): number analyzed (Participants) | 24
  Week 52 (APOE4 E4 homozygotes) | 4.2 (14.19)
  Week 24 (APOE4 E4 heterozygotes): number analyzed (Participants) | 377
  Week 24 (APOE4 E4 heterozygotes) | 1.6 (8.45)
  Week 52 (APOE4 E4 heterozygotes): number analyzed (Participants) | 82
  Week 52 (APOE4 E4 heterozygotes) | 3.7 (12.34)

ADVERSE EVENTS:
Time Frame: Up to 76 Weeks
Description: All subject (Full population) was used for analysis.
Arm/Group | RSG XR
All-Cause Mortality (participants affected / at risk) | 20/1461
Serious Adverse Events (participants affected / at risk) | 126/1461
Other Adverse Events (participants affected / at risk) | 130/1461
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSG XR (N=1461)
Fall (Injury, poisoning and procedural complications) | 4
Femur fracture (Injury, poisoning and procedural complications) | 3
Humerus fracture (Injury, poisoning and procedural complications) | 2
Skin laceration (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Drug toxicity (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Pacemaker complication (Injury, poisoning and procedural complications) | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Cerebrovascular accident (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 4
Dementia (Nervous system disorders) | 2
Dementia Alzheimer's type (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Nerve root compression (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Thalamic infarction (Nervous system disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 5
Bronchopneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paget's disease of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Refractory anaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aggression (Psychiatric disorders) | 3
Delirium (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 1
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Panic disorder (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Lumbar hernia (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1
Death (General disorders) | 1
General physical health deterioration (General disorders) | 1
Oedema peripheral (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Circulatory collapse (Vascular disorders) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1
Post thrombotic syndrome (Vascular disorders) | 1
Blood sodium increased (Investigations) | 1
Weight increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RSG XR (N=1461)
Oedema peripheral (General disorders) | 130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.